CLINICAL TRIAL: NCT00978627
Title: NN5401-3594: A 26-week, Open-labelled, Two-arm, Parallel, Randomised Trial Comparing Efficacy and Safety of NN5401 Once Daily Plus Insulin Aspart vs. Basal-bolus Treatment With Insulin Detemir Plus Insulin Aspart in Subjects With Type 1 Diabetes / NN5401-3645: An Extension Trial Comparing Safety and Efficacy of NN5401 Plus Meal-time Insulin Aspart for the Remaining Meals With Insulin Detemir Plus Meal-time Insulin Aspart in Type 1 Diabetes (BOOST™: T1)
Brief Title: Comparison of NN5401 Plus Insulin Aspart With Insulin Detemir Plus Insulin Aspart in Type 1 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3594; 2008-005769-71 (EudraCT Number); U1111-1111-8943 (Other: WHO); 2009-013412-13 (EudraCT Number); U1111-1113-2475 (Other: WHO); NCT01087606 (obsolete NCT alias)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp OD (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: insulin aspart
- IDet (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Injected subcutaneously (under the skin) once daily with a meal. Dose was individually adjusted.
  Arms: IDegAsp OD
Drug: insulin detemir — Injected subcutaneously (under the skin) once daily or twice daily. Dose was individually adjusted.
  Arms: IDet
Drug: insulin aspart — Injected subcutaneously (under the skin) at the remaining meals. Dose was individually adjusted.
  Arms: IDegAsp OD
Drug: insulin aspart — Injected subcutaneously (under the skin) as meal time insulin. Dose was individually adjusted.
  Arms: IDet

SUMMARY:
This trial is conducted in Europe, Oceania, and the United States of America (USA).

The aim of this clinical trial is to compare NN5401 (insulin degludec/insulin aspart (IDegAsp)) with insulin detemir (IDet) plus insulin aspart in patients with type 1 diabetes (main period) followed by the extension period comparing the long-term safety of NN5401 plus insulin aspart with insulin detemir plus insulin aspart.

The main period is registered internally at Novo Nordisk as NN5401-3594 while the extension period is registered as NN5401-3645.

ELIGIBILITY:
Inclusion Criteria:

* FOR THE MAIN TRIAL, NN5401-3594:
* Type 1 diabetes mellitus for at least 12 months
* Ongoing daily treatment with insulin (in a basal bolus regimen, premix insulin regimen, self mix regimen) for at least 12 months
* HbA1c 7.0-10.0% (both inclusive)
* BMI (Body Mass Index) below or equal to 35.0 kg/m^2
* FOR THE EXTENSION TRIAL, NN5401-3645:
* The subject must have completed the six-month treatment period in trial NN5401-3594

Exclusion Criteria:

* FOR THE MAIN TRIAL, NN5401-3594:
* Treatment with other insulin regimens than insulin in a basal bolus regimen/premix insulin regimen/self mix regimen within 3 months
* Cardiovascular disease within the last 6 months
* Uncontrolled treated/untreated severe hypertension
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer
* FOR THE EXTENSION TRIAL, NN5401-3645:
* Anticipated significant lifestyle changes during the trial
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (74):
- United States (28):
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, Salinas, California
  - Novo Nordisk Investigational Site, Valencia, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Eagan, Minnesota
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Seattle, Washington
- Australia (7):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Fitzroy
  - Novo Nordisk Investigational Site, Geelong
- Denmark (3):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Gentofte Municipality
- France (4):
  - Novo Nordisk Investigational Site, Auxerre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Pointe à Pitre
- Israel (3):
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Poland (4):
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Sopot
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
- Novo Nordisk Investigational Site, Bayamón, Puerto Rico
- Romania (7):
  - Novo Nordisk Investigational Site, Brasov, Brașov County
  - Novo Nordisk Investigational Site, Buzău, Buzău
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Iași
  - Novo Nordisk Investigational Site, Oradea
  - Novo Nordisk Investigational Site, Sibiu
- Russia (9):
  - Novo Nordisk Investigational Site, Kemerovo
  - Novo Nordisk Investigational Site, Kursk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Volgograd
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- [Background] Hirsch IB, Franek E, Mersebach H, Bardtrum L, Hermansen K. Safety and efficacy of insulin degludec/insulin aspart with bolus mealtime insulin aspart compared with standard basal-bolus treatment in people with Type 1 diabetes: 1-year results from a randomized clinical trial (BOOST(R) T1). Diabet Med. 2017 Feb;34(2):167-173. doi: 10.1111/dme.13068. Epub 2016 Feb 19. PMID 26773446
- [Result] Hirsch IB, Bode B, Courreges JP, Dykiel P, Franek E, Hermansen K, King A, Mersebach H, Davies M. Insulin degludec/insulin aspart administered once daily at any meal, with insulin aspart at other meals versus a standard basal-bolus regimen in patients with type 1 diabetes: a 26-week, phase 3, randomized, open-label, treat-to-target trial. Diabetes Care. 2012 Nov;35(11):2174-81. doi: 10.2337/dc11-2503. Epub 2012 Aug 28. PMID 22933438
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 79 sites in 9 countries: Denmark (3 sites), Poland (6 sites), Romania (8 sites), France (3 sites), United Kingdom (8 sites), Russian Federation (11 sites), Israel (4 sites), Australia (7 sites), and United States (29 sites). Some sites did not enrol subjects in the extension period.
Pre-assignment Details: The total duration of treatment was up to 52 weeks (26 weeks [main trial: NN5401-3594, NCT00978627] + 26 weeks [extension trial: NN5401-3645]), separated by 1 week of wash-out period; during which subjects were treated with Neutral Protamine Hagedorn (NPH) insulin twice daily (BID) in combination with insulin aspart.
Groups:
- IDegAsp OD: Insulin degludec/insulin aspart (IDegAsp) was given subcutaneously (s.c.) once daily (OD) with a main meal in combination with mealtime insulin aspart (IAsp) for the remaining meals. The regimen was given for 26 weeks in the main period and for an additional 26 weeks in the extension period.
- IDet: Insulin detemir (Idet) was given subcutaneously (s.c) once daily (OD) in the evening or twice daily (BID) in combination with mealtime insulin aspart (Iasp). The regimen was given for 26 weeks in the main period and for an additional 26 weeks in the extension period.
Period: Main: Week 0 to 26 (NN5401-3594)
Arm/Group | IDegAsp OD | IDet
Started | 366 | 182
Exposed | 362 (Four subjects withdrew prior to exposure to trial products) | 180 (Two subjects withdrew prior to exposure to trial products)
Completed | 320 | 156
Not Completed | 46 | 26
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 8 | 6
Not completed — Withdrawal criteria | 7 | 5
Not completed — Unclassified | 25 | 12
Period: Extension: Week 27 to 52 (NN5401-3645)
Arm/Group | IDegAsp OD | IDet
Started | 254 (Sixty six subjects from main trial did not continue into extension trial) | 122 (Thirty four subjects from main trial did not continue into extension trial)
Completed | 233 | 113
Not Completed | 21 | 9
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal criteria | 2 | 1
Not completed — Unclassified | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp OD | IDet | Total
Number analyzed (Participants) | 366 | 182 | 548
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.8) | 42.6 (13.8) | 41.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 100 | 276
  Male | 190 | 82 | 272
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.3 (0.7) | 8.3 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.3 (4.7) | 11.0 (4.8) | 10.5 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 26 Weeks of Treatment
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 366 | 182
percentage of glycosylated haemoglobin | -0.73 (0.83) | -0.68 (0.77)

2. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 362 | 180
Episodes/100 years of patient exposure | 3917 | 4434

3. Secondary Outcome: Main Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 26
Description: Overall mean of 9-point SMPG at 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). For 22 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 349 | 177
mmol/L | 8.0 (2.2) | 8.4 (2.5)

4. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Week 0, Week 53
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 366 | 182
percentage of glycosylated haemoglobin | -0.65 (0.81) | -0.56 (0.80)

5. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol /L.
Time Frame: Week 0 to Week 53 + 7 days follow up
Population: as for outcome 2
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 362 | 180
Episodes/100 years of patient exposure | 3183 | 3673

6. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 53 + 7 days follow up
Population: as for outcome 2
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 362 | 180
Episodes/100 years of patient exposure | 309 | 541

7. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: as for outcome 6
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: as for outcome 2
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 362 | 180
Episodes/100 years of patient exposure | 371 | 572

8. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Fasting Plasma Glucose (FPG) After 52 Weeks of Treatment
Description: Change from baseline in FPG after 52 weeks of treatment.
Time Frame: Week 0, Week 53
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). For 2 subjects, FPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 365 | 181
mmol/L | -1.83 (5.69) | -2.40 (5.86)

9. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 53 + 7 days of follow up
Population: as for outcome 2
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDegAsp OD | IDet
Number analyzed (Participants) | 362 | 180
Events/100 years of patient exposure
  Adverse event (AE) | 408 | 442
  Serious AE | 24 | 19
  Severe AE | 33 | 48
  Moderate AE | 93 | 83
  Mild AE | 282 | 311
  Fatal AE | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 to Week 53 + 7 days of follow up.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp OD | IDet
Serious Adverse Events (participants affected / at risk) | 46/362 | 20/180
Other Adverse Events (participants affected / at risk) | 166/362 | 90/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=362) | IDet (N=180)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 15 (25) | 9 (9)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Victim of crime (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=362) | IDet (N=180)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 12 (12)
Nausea (Gastrointestinal disorders) | 14 (24) | 9 (10)
Injection site reaction (General disorders) | 5 (8) | 9 (36)
Gastroenteritis (Infections and infestations) | 14 (15) | 9 (10)
Influenza (Infections and infestations) | 25 (25) | 9 (12)
Nasopharyngitis (Infections and infestations) | 89 (139) | 38 (62)
Upper respiratory tract infection (Infections and infestations) | 33 (48) | 20 (30)
Hypoglycaemia (Metabolism and nutrition disorders) | 29 (40) | 24 (50)
Headache (Nervous system disorders) | 35 (102) | 16 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.